CLINICAL TRIAL: NCT06165263
Title: The Effect of the Mobile Earthquake Education Application Developed for High School Students on Students' Knowledge Levels About Earthquakes
Brief Title: The Effect of a Mobile Earthquake Education Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Kamil Kocak, PhD Student, Principal Investigator, Dokuz Eylul University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 7586-GOA, 2022/35-19; TSA-2023-3231 (Other Grant/Funding Number: Dokuz Eylül Üniversitesi BAP)
Record Dates: First submitted 2023-12-02; First posted 2023-12-11 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2023-12

CONDITIONS: Students; Earthquake; Education
Keywords: Disaster management; disaster education; mobile application; risk management; earthquake

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): The researcher will present 2 hours of basic earthquake education to control group.
  The control group will not receive any other intervention. Control group will consist of 80 students.
- Mobile earthquake education (Experimental): The researcher will present 2 hours of basic earthquake education to experimental group.
  The students in the experimental group will use "mobile earthquake education" for 4 weeks.
  İnterventional group will consist of 80 students.
  Interventions: Behavioral: Mobile earthquake education

INTERVENTIONS:
Behavioral: Mobile earthquake education — The mobile earthquake education application was developed to increase high school students' knowledge about earthquakes through videos, activities or games. In the mobile earthquake education application, there are 4 modules that provide general information about the earthquake and what to do before, during and after the earthquake.
  Arms: Mobile earthquake education

SUMMARY:
This research aims to experimentally explore the effect of the mobile earthquake education application developed for high school students on the earthquake knowledge level and earthquake risk perception of high school students.

DETAILED DESCRIPTION:
Earthquake is the type of natural hazard with the highest mortality in the world and in Turkey. The majority of Turkey's population lives under the threat of earthquakes.It is necessary to adopt a risk management approach against earthquake danger and to raise conscious individuals.Thanks to earthquake education activities for students, earthquake awareness can be spread to students' peers, families and teachers. In this way, the society can be resistant to the earthquake hazard.It is recommended that a combination of visual, audio and interactive tools be preferred and technology be used in earthquake education activities.In earthquake education activities, the use of mobile learning method has advantages such as eliminating time and space limitations, increasing equality of opportunity in education, supporting individualized learning and providing instant feedback.

This project will be carried out to examine the effect of the mobile earthquake education application developed for high school students on the students' level of knowledge about earthquakes. The research will be conducted in two different schools in Konya in the 2023-2024 academic year.The population of the research is 9th grade students in both schools. The sample size was calculated with the Open epi and t was decided to 160 students, 80 experimental and 80 control. In order to prevent interaction between students, one of the schools involved in the research will be the experimental group and the other will be the control group. Groups will be determined with the lottery method.Three 9th grade students from each school will be included in the research. Three classes to be taken into groups in schools will be selected by simple random sampling method. The researcher will collect the pre-tests to all students who meet the research criteria and agree to participate in the study. The researcher will present 2 hours of basic earthquake education to both the experimental and control groups. The students in the experimental group will be registered on the mobile earthquake education. The students in the experimental group will use "mobile earthquake education" for 4 weeks. After 4 weeks, a posttest will be administered to all students in the experimental and control groups. To evaluate the permanence of the mobile earthquake education initiative, a post-test will be administered to participants 8 weeks after the application begins. As data collection form, sociodemographic characteristics survey form, earthquake risk perception scale, earthquake knowledge level survey will be used. The results will be presented with frequency distributions and mean±standard deviation. In the analysis, t test or Mann Whitney U Analysis will be used in independent groups and Variance Analysis or Friedman Analysis of Variance will be used in dependent groups.

ELIGIBILITY:
Inclusion Criteria:

* Being a 9th grade student in high school
* The student or parent must have an Android phone
* The student has internet access

Exclusion Criteria:

• Student's participation in any earthquake-related education

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 160 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-09-08 (Actual)

PRIMARY OUTCOMES:
Level of knowledge about earthquakes | Baseline, 4 weeks after intervention and 8 weeks after intervention .
  "Earthquake knowledge level form" will be used to determine the level of knowledge about earthquakes. It was developed in line with the literature to determine the level of knowledge about earthquakes. The form consists of 25 items containing information about the earthquake and precautions to be taken before, during and after the earthquake. Each correct answer is scored as 1 and an incorrect answer is scored as 0. The minimum score is 0 and the maximum score is 25. As the score obtained from the scale increases, the level of earthquake knowledge increases. The validity of the items in the survey form was evaluated by consulting the expert opinions of 7 academicians who work in this field.

SECONDARY OUTCOMES:
Earthquake risk perception | Baseline, 4 weeks after intervention and 8 weeks after intervention .
  "Earthquake risk perception scale" will be used to determine earthquake risk perception. The scale consists of two subscales (cognitive and emotional earthquake risk perception) and 8 items. Scoring of these items; 5 points if strongly agree, 4 points if agree, 3 points if moderately agree, 2 points if disagree and 1 point if strongly disagree. From the 5-point Likert type scale, the maximum score is 40 points and the minimum score is 8 points. An increase in the score indicates an increase in risk perception.

CONTACTS AND LOCATIONS:
Overall Officials: Kamil Koçak, PhD Student, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: 6 mounts later
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/